CLINICAL TRIAL: NCT06043791
Title: Applicability of 3T Shoulder MRI in Detection of Labral Pathology
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Courtney Scher, Orthopedic Surgeon, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16459
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Labral Tear, Glenoid
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Patients will be imaged with standard of care MRI shoulder arthrogram on a 1.5 T magnet and additionally with non-contrast MRI of the shoulder on a 3 T magnet. All patients will be dually imaged. Initial imaging will utilize the standard of care, and, subsequently, patients will be brought back within 2 weeks, for non-contrast MRI as part of the study protocol
  Interventions: Radiation: 1.5 Tesla magnet MR arthrography; Radiation: 3 Tesla magnet non-contrast MRI

INTERVENTIONS:
Radiation: 1.5 Tesla magnet MR arthrography — MR arthrogram is an invasive procedure where the patient's joint is injected with a mixture of dilute gadolinium, iodinated contrast medium, local anesthetic, and saline solution followed by imaging with 1.5 Tesla MRI.
  Other Names: MRI Arthrogram
Radiation: 3 Tesla magnet non-contrast MRI — 3T MRI uses very powerful magnets that produce a 3-tesla magnetic field. A 3-tesla magnetic field is twice as powerful as the fields used in conventional high-field MRI scanners, and as much as 15 times stronger than low-field or open MRI scanners. This results in a clearer and more complete image. Studies have shown that it is highly sensitive and specific in detecting labral and cartilage pathology

SUMMARY:
The purpose of this observational study is to compare image quality between 3 Tesla magnet (3T) non-contrast MRI to the current standard of MR arthrogram (1.5T magnet) in detecting shoulder labral and cartilage pathology.

An orthopedic surgeon on the research team will screen for patients with high probability of labral and/or cartilaginous pathology and the need for advanced imaging. The orthopedic surgeon's inclusion of patients will be based on a thorough clinical exam and obtained history. Patients included in the study will be imaged using both protocols - the current standard of MR arthrogram with a 1.5T magnet and non-contrast imaging with a 3T magnet. Both sets of images will be interpreted by multiple fellowship-trained musculoskeletal radiologists for adequate intra and inter-rater reliability.

DETAILED DESCRIPTION:
The specific aim of this investigation is to determine the accuracy and reliability of 3T MRI in the detection of shoulder labral and cartilage pathology as compared to the current standard of MR arthrography with a 1.5T magnet scanner.

Patients who present to a Henry Ford orthopedic clinic associated with a surgeon participating in this study and are indicated for labral surgery will be assessed for eligibility. Patients will be interviewed, and their medical chart reviewed to determine whether they meet inclusion and exclusion criteria. Sections of the medical chart that will be reviewed include history of present illness, medical and surgical history, and the physical exam. Patients who meet criteria for this study will be consented by the surgeon or other key study personnel. A password-protected spreadsheet stored on Henry Ford OneDrive will be used to track patients enrolled in the study and make record of patients who do not meet inclusion criteria.

Patients between 14-65 years of age being seen in orthopedic clinic with shoulder pathology likely requiring surgical intervention will be screened into the study. Patients will be imaged with standard of care MRI shoulder arthrogram on a 1.5 T magnet and additionally with non-contrast MRI of the shoulder on a 3 T magnet. All patients will be dually imaged. Initial imaging will utilize the standard of care, and, subsequently, patients will be brought back within 2 weeks, for non-contrast MRI as part of the study protocol. Both sets of images will be interpreted by multiple fellowship-trained musculoskeletal radiologists for adequate intra and inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for likely labral surgery
* Chronic, degenerative labral and/or cartilage pathology
* Ability to read and understand English
* Age ≥ 18 years
* Age ≤ 65 years

Exclusion Criteria:

* Patient does not complete both the MR arthrogram and 3T non-contrast MRI
* Unexpected trauma in between the MR arthrogram and 3T non-contrast MRI
* Age < 18 years
* Age > 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Quantitative Assessment of Labral Tear Detection: 3T Non-contrast MRI vs. MRA | 1 week
  Consistent diagnosis of labral tear in both imaging modalities done by fellowship-trained radiologists

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Muh, MD, Principal Investigator — Henry Ford Health; Courtney Scher, MD, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Health, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No